CLINICAL TRIAL: NCT02052531
Title: A Phase II, Single Center, Double-blind, Randomized Clinical Trial to Evaluate the Efficacy and Safety of PAC-14028 Cream in Dermal Pruritus
Brief Title: Evaluation of the Antipruritic Effect of PAC-14028 Cream in Skin Pruritus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-TRPV1_PII-01
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Skin Pruritus
MeSH Terms: interventions — N-(1-(3,5-difluoro-4-methanesulfonylaminophenyl)ethyl)-3-(2-propyl-6-trifluoromethylpyridine-3-yl)acrylamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PAC-14028 cream 0.3% (Experimental): PAC-14028 cream 0.3%, twice daily for 28 days
  Interventions: Drug: PAC-14028
- PAC-14028 cream 1.0% (Experimental): PAC-14028 cream 1.0%, twice daily for 28days
  Interventions: Drug: PAC-14028
- Vehicle (Placebo Comparator): Vehicle, twice daily for 28days
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: PAC-14028 — Participants received topical PAC-14028 cream 0.3 or 1% twice daily for 4 weeks
  Other Names: PAC-14028 Cream 0.3%; PAC-14028 Cream 1.0%
  Arms: PAC-14028 cream 0.3%; PAC-14028 cream 1.0%
Other: Vehicle — Participants received topical Vehicle twice daily for 4 weeks
  Other Names: Vehicle of PAC-14028 Cream
  Arms: Vehicle

SUMMARY:
The objective of this study was to find a clinically appropriate dose of PAC-14028 cream by comparatively evaluating the efficacy and safety of PAC-14028 cream of Amorepacific Corporation in patients with dermal pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at the age of 20 to 65 years old (both inclusive)
* Pruritus test ≥ 5cm (10cm Visual Analogue Scale [VAS]) at baseline
* Eczema or dry skin on the study drug application site
* Women of childbearing potential should have a negative urine pregnancy test at screening and agree to employ an effective method of birth control (surgical sterilization or oral contraceptives, barrier method with spermicides, intrauterine device, etc.) during the study period.
* Voluntarily signed written informed consent forms for study participation.

Exclusion Criteria:

* Pruritus due to other medical (liver disease, renal failure, etc.), psychotic, or neuropathic causes rather than as a skin disease.
* Chronic skin diseases such as malignant tumor or chronic urticaria, among skin diseases.
* Simple pruritus caused by allergic substances such as scabies or insect bites.
* Presence of symptoms of generalized infection at the time of study participation.
* Previous local treatment or antibiotics administration for pruritus within 7 days prior to study participation.
* Previous use of oral steroids within 1 month and local steroids within 2 weeks prior to study participation.
* History of physical treatment for pruritus, including phototherapy, within 1 month prior to study participation.
* Patients who are treated with prohibited concomitant drugs or considered to inevitably require treatment with prohibited concomitant drugs during the study period.
* Renal function impairment with creatinine level
* Hepatic function impairment with aspartate aminotransferase (AST)/ alanine aminotransferase (ALT)
* Pregnant and lactating women
* Participation in another clinical study within 1 month prior to screening.
* Patients considered ineligible for study participation by the principal investigator or sub-investigator for other reasons; pruritus due to other medical (liver disease, renal failure, etc.), psychotic, or neuropathic causes rather than as a skin disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) | Baseline through Study Day 28
  Patient reported outcome of pruritis measurement on a change in visual analog scale

SECONDARY OUTCOMES:
Treatment success rate | Baseline through Study Day 28
Change in specified symptom sum score (SRRC) Index | Baseline through Study Day 28
Change in transepidermal water loss | Baseline through Study Day 28
Change in skin hydration | Baseline through Study Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Han Kim, MD,Ph.D, Principal Investigator — Department of Dermatology, Seoul National University Hospital
Locations (1):
- Kyu-Han Kim, Seoul, South Korea